CLINICAL TRIAL: NCT01396187
Title: A Phase 1, Placebo-Controlled Randomized Trial To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Ascending Intravenous Doses Of PF-05231023 In Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Tolerability of Ascending Intravenous Doses of PF-05231023 In Adult Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2901002
Record Dates: First submitted 2011-07-06; First posted 2011-07-18 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; safety; multiple dose; intravenous
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-05231023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: PF-05231023
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-05231023 — 5 mg IV twice a week for 4 weeks
  Arms: Treatment
Drug: PF-05231023 — 25 mg IV twice a week for 4 weeks
  Arms: Treatment
Drug: PF-05231023 — 100 mg IV twice a week for 4 weeks
  Arms: Treatment
Drug: PF-05231023 — 200 mg IV twice a week for 4 weeks
  Arms: Treatment
Other: Placebo — 0.9% w/v sodium chloride injection, United States Pharmacopeia (USP), twice a week IV for 4 weeks
  Arms: Placebo

SUMMARY:
This is a trial in subjects with Type 2 diabetes mellitus to study the safety, tolerability and pharmacokinetics of multiple ascending doses of PF-05231023.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and female subjects of non-childbearing potential between the ages of 30 and 70 years, inclusive, with a historical diagnosis of type 2 diabetes mellitus, diagnosed according to the American Diabetes Association guidelines. Subjects who have other conditions but are well controlled by either diet or medications may be included as well (for example, a subject with high cholesterol level on appropriate treatment is eligible).
* Body Mass Index (BMI) of 25 to 35.5 kg/m2, and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Diagnosis of Type 1 diabetes mellitus.
* Evidence of diabetic complications with significant end organ damage

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2901002&StudyName=Safety%20and%20Tolerability%20of%20Ascending%20Intravenous%20Doses%20of%20PF-05231023%20In%20Adult%20Subjects%20with%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a historical diagnosis of type 2 diabetes mellitus (T2DM), diagnosed according to the American Diabetes Association (ADA) guidelines, those with well controlled diabetes and were on stable metformin therapy were recruited in the study.
Pre-assignment Details: Dose of PF-05231023 was escalated based on sponsor's and investigator's discretion, depending upon safety, tolerability and pharmacokinetic profile of PF-05231023.
Groups:
- Placebo: Placebo matched to PF-05231023 intravenous infusion over approximately 1 hour on Day 1, 4, 8, 11, 15, 18, 22 and 25.
- PF-05231023 5 mg: PF-05231023 5 mg (milligram) intravenous infusion over approximately 1 hour on Day 1, 4, 8, 11, 15, 18, 22 and 25.
- PF-05231023 25 mg: PF-05231023 25 mg intravenous infusion over approximately 1 hour on Day 1, 4, 8 11, 15, 18, 22 and 25.
- PF-05231023 100 mg: PF-05231023 100 mg intravenous infusion over approximately 1 hour on Day 1, 4, 8, 11, 15, 18, 22 and 25.
- PF-05231023 140 mg: PF-05231023 140 mg intravenous infusion over approximately 1 hour on Day 1, 4, 8, 11, 15, 18, 22 and 25.
Period: Overall Study
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Started | 8 | 12 | 10 | 10 | 10
Completed | 7 | 9 | 9 | 10 | 9
Not Completed | 1 | 3 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Groups:
- PF-05231023 5 mg: PF-05231023 5 mg intravenous infusion over approximately 1 hour on Day 1, 4, 8, 11, 15, 18, 22 and 25.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg | Total
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (4.3) | 50.2 (10.0) | 56.9 (6.9) | 59.0 (6.3) | 57.6 (9.1) | 55.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 3 | 4 | 11
  Male | 6 | 11 | 9 | 7 | 6 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included assessment of height, weight, blood pressure, pulse rate and body temperature. Criteria for abnormal physical findings was based on investigator's discretion and were reported as adverse event (AE), as planned.
Time Frame: Baseline up to Day 42
Population: Physical examination data reported in this study was for identification of adverse events and were reported as adverse event in the AE section.
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 77 which were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Day 77
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10
participants
  AEs | 5 | 6 | 3 | 8 | 10
  SAEs | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (RBCs)(less than [<] 0.8*lower limit of normal[LLN]); leucocytes (<0.6/greater than [>]1.5*upper limit of normal [ULN]); platelets (<0.5*LLN></0>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN></0>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin, direct bilirubin, indirect bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN></0>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN></0>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN></0>1.1*ULN); urine RBCs, urine white blood cells (WBCs) (> or equal[=]20 high-powered field), urine bacteria >20 high-powered field. Total number of participants with any laboratory abnormalities were reported.
Time Frame: Baseline up to Day 42
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10
participants | 8 | 10 | 9 | 9 | 10

4. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for vital signs abnormalities: supine systolic blood pressure (SBP) <90 millimeter of mercury (mm Hg), supine diastolic BP (DBP) <50 mm Hg, supine pulse rate <40 beats per minute (bpm), > 120 bpm. Maximum increase or decrease from baseline in supine SBP >=30 mm Hg and maximum increase or decrease from baseline in supine DBP >=20 mm Hg.
Time Frame: Baseline up to Day 77
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10
participants
  SBP < 90 mm Hg | 0 | 0 | 2 | 0 | 1
  DBP< 50 mm Hg | 0 | 0 | 0 | 0 | 0
  Pulse rate < 40 bpm | 0 | 0 | 0 | 0 | 0
  Pulse rate > 120 bpm | 0 | 0 | 0 | 0 | 0
  SBP: Maximum increase >= 30 mm Hg | 3 | 1 | 3 | 2 | 0
  DBP: Maximum increase >=20 mm Hg | 1 | 1 | 1 | 1 | 1
  SBP: Maximum decrease>=30 mm Hg | 2 | 0 | 0 | 1 | 3
  DBP: Maximum Decrease >= 20 mm Hg | 1 | 0 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for potential clinical concern in ECG parameters: maximum PR interval of greater than or equal to (>=) 300 milliseconds (msec), maximum QRS interval >=140 msec, maximum QTCF interval (Fridericia's Correction) of 450 to <480 msec, 480 to <500 msec and >=500 msec, maximum increase of >=25 percent (%) for baseline value of >200 msec and >=50% for baseline value of less than or equal to (<=) 200 msec for PR interval, maximum increase from baseline of >=50% for QRS interval, maximum increase from baseline of >=30 msec to <60 msec and maximum increase from baseline of >60 msec in QTCF interval (Fridericia's Correction).
Time Frame: Baseline up to Day 77
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10
participants
  Maximum PR interval >=300 msec | 0 | 0 | 0 | 0 | 0
  Maximum QRS Complex >=140 msec | 0 | 0 | 0 | 0 | 0
  Maximum QTCF interval 450 to <480 msec | 0 | 0 | 0 | 0 | 2
  Maximum QTCF interval 480 to <500 msec | 0 | 0 | 0 | 0 | 0
  Maximum QTCF interval >=500 msec | 0 | 0 | 0 | 0 | 0
  PR interval increase from baseline >=25/50% | 0 | 0 | 0 | 0 | 0
  QRS complex increase from baseline >=50% | 0 | 0 | 0 | 0 | 0
  QTCF interval increase from baseline 30 to <60msec | 1 | 1 | 1 | 0 | 1
  QTCF interval increase from baseline >=60 msec | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Blood Glucose Abnormalities
Description: Criteria for blood glucose abnormality: Blood glucose levels <0.6* LLN or >1.5* ULN.
Time Frame: Baseline up to Day 32
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 10
participants
  <0.6*LLN | 0 | 0 | 0 | 0 | 0
  >1.5*ULN | 6 | 6 | 6 | 5 | 9

7. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-05231023 After Single Dose
Description: Participants who received PF-05231023 with C-terminal and N-terminal AUCtau were reported.
Time Frame: 0 hour (pre-dose) on Day 1, 4; 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 1; Day 2, 3
Population: Pharmacokinetic (PK) parameter analysis set included all enrolled and treated participants who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 12 | 10 | 10 | 10
nanogram*hour per milliliter (ng*hr/mL)
  C-terminal | 12680 (23) | 58780 (23) | 229500 (22) | 365300 (22)
  N- terminal | 33240 (22) | 186800 (16) | 844200 (12) | 1051000 (19)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05231023 After Single Dose
Description: Participants who received PF-05231023 with C-terminal and N-terminal Tmax were reported.
Time Frame: as for outcome 7
Population: PK parameter analysis set included all enrolled and treated participants who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 12 | 10 | 10 | 10
hour
  C- terminal | 1.02 [0.500 to 1.50] | 1.26 [1.00 to 2.00] | 1.25 [0.883 to 2.00] | 1.50 [1.00 to 2.15]
  N-terminal | 1.50 [0.500 to 2.00] | 1.50 [1.02 to 5.00] | 1.50 [1.00 to 2.97] | 1.50 [1.07 to 5.00]

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05231023 After Single Dose
Description: Participants who received PF 05231023 with C-terminal and N-terminal Cmax were reported.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 12 | 10 | 10 | 10
nanogram per milliliter (ng/mL)
  C -terminal | 1270 (11) | 5991 (17) | 23500 (21) | 34390 (15)
  N -terminal | 1182 (18) | 7123 (18) | 28480 (18) | 35790 (17)

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-05231023 at Steady State
Description: Participants who received PF-05231023 with C-terminal and N-terminal AUCtau at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: PK parameter analysis set included all enrolled and treated participants who had at least 1 of the PK parameters of interest. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ng*hr/mL
  C-terminal | 14810 (33) | 73940 (27) | 324300 (15) | 453400 (21)
  N-terminal | 65420 (16) | 317800 (11) | 1533000 (24) | 1990000 (22)

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-05231023 at Steady State
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) at steady state. Participants who received PF-05231023 with C-terminal and N-terminal AUClast at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ng*hr/mL
  C-terminal | 11280 (26) | 52710 (23) | 294100 (26) | 456700 (21)
  N-terminal | 121900 (27) | 590400 (11) | 2859000 (20) | 3196000 (25)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05231023 at Steady State
Description: Participants who received PF-05231023 with C-terminal and N-terminal Tmax at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
hour
  C-terminal | 1.42 [1.02 to 1.48] | 1.48 [1.00 to 2.00] | 1.40 [1.00 to 3.00] | 1.01 [1.00 to 1.50]
  N-terminal | 1.48 [1.42 to 1.48] | 1.45 [0.500 to 13.0] | 1.99 [1.37 to 24.0] | 1.45 [1.00 to 2.00]

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05231023 at Steady State
Description: Participants who received PF 05231023 with C-terminal and N-terminal Cmax at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ng/mL
  C-terminal | 1239 (23) | 5629 (21) | 27240 (16) | 37160 (13)
  N-terminal | 1839 (21) | 9016 (17) | 37770 (18) | 61160 (16)

14. Secondary Outcome: Accumulation Ratio for Area Under the Curve From Time Zero to End of Dosing Interval of PF-05231023 (Rac)
Description: Rac was obtained from AUCtau at steady state (Day 25) divided by AUCtau after single dose (Day 1). AUCtau was the area under the concentration-time profile from time zero to end of dosing interval, where tau = 72 hours for Day 1 and tau = 96 hours for Day 25. Participants who received PF-05231023 with C-terminal and N-terminal Rac at steady state were reported.
Time Frame: 0 hour (pre-dose) on Day 1, 4, 25; 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 1, 25; Day 2, 3, 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ratio
  C-terminal | 1.258 (20) | 1.258 (24) | 1.413 (10) | 1.173 (8)
  N-terminal | 2.016 (18) | 1.702 (15) | 1.818 (24) | 1.810 (14)

15. Secondary Outcome: Accumulation Ratio for Maximum Observed Plasma Concentration (Rac,Cmax) of PF- 05231023
Description: Accumulation ratio based on maximum plasma concentration (Cmax) was calculated as: Rac,Cmax = Cmax at steady state (Day 25) divided by Cmax at first dose (Day 1). Participants who received PF-05231023 with C-terminal and N-terminal Rac,Cmax at steady state were reported.
Time Frame: as for outcome 14
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ratio
  C-terminal | 0.9992 (19) | 0.9392 (20) | 1.159 (13) | 1.033 (12)
  N-terminal | 1.626 (17) | 1.266 (23) | 1.326 (19) | 1.642 (8)

16. Secondary Outcome: Plasma Terminal Half-Life (t1/2) of PF-05231023 at Steady State
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half at the terminal phase. Participants who received PF-05231023 with C-terminal and N-terminal t1/2 at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: PK parameter analysis set included all enrolled and treated participants who had at least 1 of the PK parameters of interest. "n" signifies those participants who were evaluated for this measure at the specified terminal for each arm.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 12 | 10 | 10 | 10
hour
  C-terminal (n=8, 7, 10, 8) | 6.484 (0.79685) | 7.879 (0.78138) | 9.563 (2.5419) | 10.25 (1.5121)
  N-terminal (n=9, 10, 9, 6) | 83.93 (10.922) | 84.38 (8.7742) | 97.47 (14.534) | 74.62 (13.781)

17. Secondary Outcome: Apparent Clearance (CL) of PF-05231023 at Steady State
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Participants who received PF-05231023 with C-terminal and N-terminal CL at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: liter per hour
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
liter per hour
  C-terminal | 0.3378 (26) | 0.3383 (23) | 0.3083 (15) | 0.3086 (23)
  N-terminal | 0.07642 (14) | 0.07871 (12) | 0.06521 (21) | 0.07043 (26)

18. Secondary Outcome: Volume of Distribution of PF-05231023 at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state. PF-05231023 with C-terminal and N-terminal Vss at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 16
Measure: Geometric Mean (Standard Deviation); unit: liter
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 12 | 10 | 10 | 10
liter
  C-terminal (n=8, 7, 10, 8) | 1.467 (19) | 1.873 (16) | 2.940 (48) | 4.110 (12)
  N-terminal (n=9, 10, 9, 6) | 7.320 (20) | 7.594 (15) | 6.570 (33) | 4.863 (18)

19. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-05231023 at Steady State
Description: Participants who received PF 05231023 with C-terminal and N-terminal Cmax at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ng/mL
  C-terminal | 0.0003894 (6.8667) | 0.1538 (11.864) | 80.51 (102) | 218.8 (76)
  N-terminal | 550.5 (33) | 1861 (30) | 9987 (21) | 12440 (29)

20. Secondary Outcome: Average Plasma Concentration (Cav) of PF-05231023 at Steady State
Description: Participants who received PF-05231023 with C-terminal and N-terminal Cmax at steady state were reported.
Time Frame: 0 hour (pre-dose) 0.5, 1 (end of infusion), 1.5, 2, 3, 5, 9, 13 hours post-start of infusion on Day 25; Day 26, 29
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Number analyzed (Participants) | 9 | 10 | 10 | 8
ng/mL
  C-terminal | 205.5 (33) | 1027 (27) | 4504 (15) | 6300 (21)
  N-terminal | 908.6 (16) | 4411 (11) | 21290 (24) | 27620 (22)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-05231023 5 mg | PF-05231023 25 mg | PF-05231023 100 mg | PF-05231023 140 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 0/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 5/8 | 6/12 | 3/10 | 8/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | PF-05231023 5 mg (N=12) | PF-05231023 25 mg (N=10) | PF-05231023 100 mg (N=10) | PF-05231023 140 mg (N=10)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | PF-05231023 5 mg (N=12) | PF-05231023 25 mg (N=10) | PF-05231023 100 mg (N=10) | PF-05231023 140 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 5 | 4
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 2
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 0 | 0 | 1 | 4
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.